CLINICAL TRIAL: NCT05694975
Title: Clinical Efficacy of Megadose Vitamin C in Severe and Critical Ill COVID-19 Patients (CEMVISCC): A Multicenter, Randomized, Single-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy of Megadose Vitamin C in Severe and Critical Ill COVID-19 Patients.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhanguo, Clinical Efficacy of Megadose Vitamin C in Severe and Critical Ill COVID-19 Patients (CEMVISCC): A Multicenter, Randomized, Single-blind, Placebo-controlled Clinical Trial, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-KY-001-02
Record Dates: First submitted 2023-01-14; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Vitamin C; COVID-19 Pneumonia
Keywords: Vitamin C; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, randomized, single-blind, placebo-controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): 12 g Vitamin C will be infused within 6 hours by an infusion pump. This treatment will be repeated every 12 hours for 4 days.
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): The control group is assigned a placebo (5% glucose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — The total dosage of vitamin C for the treatment group is 24 g per day.
  Arms: Vitamin C
Drug: Placebo — The total dosage of placebo(5% glucose) for the control group is 24 g per day.
  Arms: Placebo

SUMMARY:
The main aim is to determine whether vitamin C can reduce 28-day all-cause mortality or persistent organ dysfunction compared with placebo in patients with severe and critical ill COVID-19 patients.

Participants will randomly receive HIVC or placebo for 4 days once enrolled. The primary outcome is a composite of death or persistent organ dysfunction (defined as dependency on vasopressors, mechanical ventilation, or CRRT) at day 28 after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18 years or older).
2. Diagnosed with COVID-19 according to the Diagnosis and Clinical Management of COVID-19. (trial version 10).
3. severe and critical ill patients with COVID-19.
4. Patients who voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients with a history of allergy to VC.
2. Pregnant or lactating women.
3. Patients with end-stage malignant tumour.
4. Patients with an expected survival duration of less than 24 hours.
5. Patients with cerebral hernia and severe craniocerebral injury.
6. Patients with diabetes.
7. Patients with a previous history of G-6-PD deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2023-01-13 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The 28-day mortality or persistent organ dysfunctionat day 28. | 28 days.
  Persistent organ dysfunction was defined as dependency on vasopressors, mechanical ventilation, or new and persisting RRT.

SECONDARY OUTCOMES:
Changes in the Sepsis-Related Organ Failure Assessment (SOFA) score. | 4 days.
  The SOFA score range from 0 (mild) to 24 (critical ill). Change = (Day 4 score - Baseline score)
Change in Plasma Inflammatory Biomarker Concentrations. | 4 days.
Changes in oxygenation index and partial pressure of carbon dioxide in arterial blood gases. | 4 days.
The duration of ventilation and vasopressor use. | 28 days.
The length of ICU stay and hospital stay. | 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Zhanguo, MD,PhD, Study Chair — Southern Medical University, China
Locations (4):
- China (4):
  - Department of Critical Care Medicine of Zhujiang Hospital, Guanzhou, Guangdong
  - Yunfu People's Hospital, Yunfu, Guangdong
  - Department of Critical Care Medicine of Zhongshan People's Hospital, Zhongshan, Guangzhou
  - the Affiliated Nanhua Hospital, Hengyang, Hunan